CLINICAL TRIAL: NCT01601756
Title: Joint Line Reconstruction in Navigated Total Knee Arthroplasty Revision
Acronym: NavRevKnie
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Aesculap AG (Industry)
Responsible Party: Principal Investigator, Georg Matziolis, Professor, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AAG-I-H-0917
Record Dates: First submitted 2012-05-14; First posted 2012-05-18 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Revision Total Knee Arthroplasty Because of; Loosening; Instability; Impingement; or Other Reasons Accepted as Indications for TKA Exchange.; The Focus is to Determine the Precision of Joint Line Restoration in Navigated vs. Conventional Revision Total Knee Arthroplasty
Keywords: revision knee arthroplasty; navigation; joint line

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- navigated revision total knee arthroplasty (Experimental): revision total knee arthroplasty with the aid of a navigation system
  Interventions: Device: navigated revision knee arthroplasty
- conventional revision knee arthroplasty (Active Comparator): revision knee arthroplasty using conventional instruments
  Interventions: Device: conventional revision knee arthroplasty

INTERVENTIONS:
Device: navigated revision knee arthroplasty — revision knee arthroplasty with the aid of a navigation system the navigation system is the Orthopilot System with a software specifically dedicated for revision operations (TKR 1.0). The system is from Aesculap AG (Tuttlingen).
  Arms: navigated revision total knee arthroplasty
Device: conventional revision knee arthroplasty — revision knee arthroplasty using conventional instruments
  Arms: conventional revision knee arthroplasty

SUMMARY:
Hypothesis: navigated revision total knee arthroplasty results in a more precise reconstruction of preoperatively planned joint line than conventional revision total knee arthroplasty (rTKA).

ELIGIBILITY:
Inclusion Criteria:

* indication for revision knee arthroplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Restoration of Joint Line | postoperatively (6 to 12 weeks after operation, we expect a mean of 9 weeks)
  Difference between preoperatively planned and postoperatively achieved joint line

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Department, Charité - University Medicine Berlin, Berlin, State of Berlin, Germany